CLINICAL TRIAL: NCT05443802
Title: Comparison of a Low Dose to a Standard Dose of Insulin in Adult Diabetic Ketoacidosis in ICU to Reduce Metabolic Complications : a Randomized, Controlled Study
Brief Title: Comparison of a Low Dose to a Standard Dose of Insulin in Adult DKA in ICU to Reduce Metabolic Complications
Acronym: LOSTINDIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP210081
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Ketoacidosis
Keywords: Diabetic ketoacidosis; Insulin deficiency; Hypoglycemia; Hypokalemia; Metabolic complications
MeSH Terms: conditions — Diabetic Ketoacidosis; Hypoglycemia; Hypokalemia | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Reduced dose of rapid-acting insulin of 0.05 IU/kg/h from randomization until resolution of DKA
  Interventions: Drug: Insulin 0.05 IU/kg/h
- Control (Other): Rapid-acting insulin dose of 0.10 IU/kg/h in accordance with usual recommendations until resolution of DKA
  Interventions: Drug: Insulin 0.10 IU/kg/h

INTERVENTIONS:
Drug: Insulin 0.05 IU/kg/h — In the experimental arm, the patients will be given an insulin dose of 0.05 IU/kg/h.
  Arms: Experimental
Drug: Insulin 0.10 IU/kg/h — In the control arm, patients will receive an insulin dose of 0.10 IU/kg/h.
  Arms: Control

SUMMARY:
Diabetic ketoacidosis (DKA), a frequent complication of diabetes, is the consequence of a profound insulin deficiency responsible for osmotic polyuria and thus major losses of water, glucose, sodium and potassium as well as a metabolic acidosis due to the uncontrolled production of ketonic acids. Management includes fluid replacement, insulin therapy and correction of metabolic disorders (including potassium loss).

Initially described in patients with type 1 diabetes (T1D), it is now often observed in patients with type 2 diabetes (T2D) in whom it is more a matter of insulin resistance than an absolute deficiency. However, international guidelines recommend a similar dose of intravenous insulin (0.10 IU/kg/hour) regardless of the type of diabetes.

During treatment, metabolic complications are frequent and potentially serious, especially in T2D due to cardiovascular comorbidities.

The research hypothesis is that decreasing the insulin dose will reduce metabolic complications without influencing time to resolution in adult patients, regardless of diabetes type.

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA), a frequent complication of diabetes, is the consequence of a profound insulin deficiency responsible for osmotic polyuria which leads to major losses of water, sodium and potassium as well as the generation of metabolic acidosis due to the uncontrolled production of ketonic acids. Management includes fluid replacement, insulin therapy and correction of metabolic disorders (including potassium loss and acidosis).

Initially described in patients with type 1 diabetes (T1D), it is now often observed in patients with type 2 diabetes (T2D) in whom it is more insulin resistance than absolute deficiency. However, international guidelines recommend a similar dosage of intravenous insulin (0.10 IU/kg/hour) regardless of the type of diabetes.

During treatment, metabolic complications are frequent and potentially serious, especially in T2D due to cardiovascular comorbidities.

A British study reported 27.6% hypoglycaemia and 55% hypokalemia during the first 24 hours of treatment. Comparable figures were observed by conducting a multicenter retrospective study of 122 patients: hypokalaemia and hypoglycaemia were observed in nearly two thirds of cases.

A pediatric study showed that a lower dose of insulin (0.05 IU/kg/h) reduced the rate of hypoglycaemia (20% vs 4%) and hypokalaemia (48% vs 20%) compared to at the standard dose (0.10 IU/kg/h) without modifying the time to resolution. But the very small number (25 children per arm), the questionable statistical analysis and the pediatric population (T1D only) do not make it possible to anticipate the potential benefit in a much more heterogeneous adult population.

The hypothesis of the research is that decreasing the insulin dose will reduce metabolic complications without influencing time to resolution in adult patients, regardless of diabetes type.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or above
* Admission in Intense/Intermediate Care Unit
* Severe DKA due to all types of diabetes (T1D, T2D and secondary diabetes and inaugural ketoacidosis) defined by association of the following 3 parameters:
* glucose > 11 mmol/L or affirmation of having diabetes
* ketonemia > 3mmol/L or ketonuria ≥ 2
* bicarbonate < 15 mmol/L and/or venous pH < or=7.3
* Randomization possible before 15UI of insulin administrated in total
* Informed and written consent. In the absence of parent/ relative/ person of trust, the patient may be included via the emergency procedure and consent will be obtained as soon as possible

Exclusion Criteria:

* Non-diabetic ketoacidosis (fasting or alcoholic)
* Patient weighing less than 30 kg
* Hypokalemia < 3.5 mmol/L at the time of inclusion
* Hyperosmolar hyperglycemic state (defined as efficient plasma osmolarity > 320 mosmol/L)
* Absence of social security coverage
* Pregnant or breastfeeding patient
* Patient under tutelage or curators
* Patient deprived of liberty due to a judicial or administrative decision
* Patient with a renal disease requiring dialysis
* Acute or chronic liver failure with Factor V < 50%
* Patient receiving a high dose of corticosteroids (≥ 0.5 mg/kg) daily
* Patient included in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Metabolic complications | 48 hours
  Proportion of patients with metabolic complications (hypokalaemia <3.5 mmol/L and/or hypoglycemia <3.9 mmol/L) treated with a reduced dose of insulin (0.05 IU/kg/h) compared with the control group receiving the 0.10 IU/kg/h dose.

SECONDARY OUTCOMES:
Resolution of diabetic ketoacidosis | 48 hours
  Time in hours between randomisation and resolution of diabetic ketoacidosis (defined by ph>7.3 and ketonemia < 3 mmol/L and bicarbonates> 15 mmol/L)
Episode of hypokalaemia | 48 hours
  Proportion of patients with at least one episode of hypokalaemia < 3.5 mmol/L between randomization and resolution of DKA
Episode of hypoglycemia | 48 hours
  Proportion of patients with at least one episode of hypoglycemia < 3.9 mmol/L between randomization and resolution of DKA
Episode of severe hypoglycemia | 48 hours
  Proportion of patients with at least one episode of hypoglycemia < 2.9 mmol/L between randomization and resolution of DKA
Cardiac arrythmia diagnosed by EKG | 48 hours
  Proportion of patients with onset of new cardiac arrhythmia diagnosed by EKG analysis (atrial fibrillation and ventricular arrhythmia) and scopic monitoring between randomization and resolution of DKA
Glucose infusion 1000mL | 48 hours
  Proportion of patients who received more than 1000 mL of 10% glucose solution (indicating tendency of hypoglycemia) between randomization and resolution of DKA or 48h after inclusion if DKA is unresolved
Glucose infusion of 30% glucose solution | 48 hours
  Proportion of patients who received one perfusion of 30% glucose solution between randomization and resolution of DKA or 48h after inclusion if DKA is unresolved
Amount of glucose perfused | 48 hours
  Amount of glucose perfused (in grams) (glucose 5%, 10% and 30%) between randomization and resolution of the DKA or 48 hours after inclusion if the DKA is not resolved
Potassium intake | 48 hours
  Potassium intake (in grams) orally and intravenously between patient randomization and resolution of DKA or 48 hours after inclusion if DKA is not resolved
Length of stay in ICU | 48 hours
  Duration of stay (in hours) in ICU
Time between patient randomization and resolution of DKA in T1D population | 48 hours
  Time in hours between patient randomization and resolution of DKA in T1D population
Time between patient randomization and resolution of DKA in T2D population | 48 hours
  Time in hours between patient randomization and resolution of DKA in T2D population
Time between patient randomization and resolution of DKA in patients suffering from first ketoacidosis episode | 48 hours
  Time in hours between patient randomization and resolution of DKA in patients suffering from ketoacidosis
Episode of hypokalaemia in T1D population | 48 hours
  Proportion of patients with at least one episode of hypokalaemia < 3.5 mmol/L between randomisation and resolution of DKA or 48 hours after inclusion if DKA is not resolved within T1D population
Episode of hypokalaemia in T2D population | 48 hours
  Proportion of patients with at least one episode of hypokalaemia < 3.5 mmol/L between randomisation and resolution of DKA or 48 hours after inclusion if DKA is not resolved within T2D population
Episode of hypokalaemia in patients suffering from first ketoacidosis episode | 48 hours
  Proportion of patients with at least one episode of hypokalaemia < 3.5 mmol/L between randomisation and resolution of DKA or 48 hours after inclusion if DKA is not resolved within inaugural ketoacidosis population
Episode of hypoglycaemia in T1D population | 48 hours
  Proportion of patients with at least one episode of hypoglycaemia < 3.9 mmol/L between randomization and resolution of DKA or 48 hours after inclusion if DKA is not resolved within T1D population
Episode of hypoglycaemia in T2D population | 48 hours
  Proportion of patients with at least one episode of hypoglycaemia < 3.9 mmol/L between randomization and resolution of DKA or 48 hours after inclusion if DKA is not resolved within T2D population
Episode of hypoglycaemia in patients suffering from first ketoacidosis episode | 48 hours
  Proportion of patients with at least one episode of hypoglycaemia < 3.9 mmol/L between randomization and resolution of DKA or 48 hours after inclusion if DKA is not resolved within inaugural ketoacidosis population
Episode of severe hypoglycaemia in T1D population | 48 hours
  Proportion of patients with at least one episode of severe hypoglycaemia < 2.9 mmol/L between randomization and resolution of DKA or 48 hours after inclusion if DKA is not resolved within T1D population
Episode of severe hypoglycaemia in T2D population | 48 hours
  Proportion of patients with at least one episode of severe hypoglycaemia < 2.9 mmol/L between randomization and resolution of DKA or 48 hours after inclusion if DKA is not resolved within T2D population
Episode of severe hypoglycaemia in patients suffering from first ketoacidosis episode | 48 hours
  Proportion of patients with at least one episode of severe hypoglycaemia < 2.9 mmol/L between randomization and resolution of DKA or 48 hours after inclusion if DKA is not resolved within inaugural ketoacidosis population

CONTACTS AND LOCATIONS:
Overall Officials: Damien Roux, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Louis Mourier Hospital, Colombes, France

IPD SHARING:
Plan to Share IPD: Undecided